CLINICAL TRIAL: NCT00003701
Title: A Phase III Randomized Trial of Either M-VAC or Paclitaxel + Carboplatin as Postoperative Adjuvant Therapy in Patients With Muscle-Invasive Transitional Cell Carcinoma of the Bladder at High-Risk for Relapse
Brief Title: Combination Chemotherapy in Treating Patients With Bladder Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066808; E-1897
Record Dates: First submitted 1999-11-01; First posted 2004-04-23 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Bladder Cancer; Urethral Cancer
Keywords: stage III bladder cancer; transitional cell carcinoma of the bladder; urethral cancer associated with invasive bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Carboplatin; Cisplatin; Doxorubicin; Methotrexate; Paclitaxel; Vinblastine

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: doxorubicin hydrochloride
Drug: methotrexate
Drug: paclitaxel
Drug: vinblastine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known whether four-drug combination chemotherapy is more effective than two-drug combination chemotherapy in treating bladder cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of two combination chemotherapy regimens in treating patients who have bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the recurrence rates and overall survival of patients treated with postoperative adjuvant methotrexate, vinblastine, doxorubicin and cisplatin (M-VAC) to those treated with combination paclitaxel and carboplatin for muscle invasive bladder cancer at particularly high risk of relapse. II. Compare the relative toxicities of postoperative M-VAC versus those encountered with postoperative paclitaxel and carboplatin. III. Compare the quality of life scores during and following completion of treatment of patients in these two treatment arms.

OUTLINE: This is a randomized study. Patients are stratified by N stage (N0 vs N+) and performance status (0-1 vs 2). Patients are randomized to receive methotrexate, vinblastine, doxorubicin, and cisplatin (arm I) or paclitaxel and carboplatin (arm II). Arm I: Patients receive methotrexate IV push on days 1, 15, and 22; vinblastine IV push on days 2, 15, and 22; doxorubicin IV push on day 2; and cisplatin IV over 2 hours on day 2. Treatment repeats every 28 days for 4 courses. Arm II: Patients receive paclitaxel IV over 3 hours on days 1 followed by carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 4 courses. Quality of life assessments are completed pretreatment, prior to course 3, 6 weeks after the last dose of chemotherapy, and at 6, 12, and 24 months from the end of therapy. Patients are followed every 3 months until year 2, every 6 months for years 2-5, and then annually thereafter.

PROJECTED ACCRUAL: There will be 490 patients accrued into this study within 2.6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed transitional cell carcinoma of the bladder or mixed histologies containing a component of transitional cell carcinoma Must have undergone radical cystectomy and pelvic lymph node dissection within 12 weeks prior to randomization No evidence of distant metastatic disease on pre- or postoperative radiographic scans No positive surgical margins in the cystectomy specimen and no known macroscopic residual disease left at time of cystectomy No bladder sparing surgery May have undergone continent urinary diversion or neobladder procedure but must have recovered completely from the effects of surgery Must have muscle-invasive disease on final pathologic staging and have a primary tumor stage of pT4, any N, M0, or any pT, N+, M0, or pT3b, any N, any M, and following a pelvic lymph node dissection have a pathologic nodal stage of pN0 (only if pT3b or pT4), pN1, or pN2 Clinically unsuspected organ confined prostate cancer found during cystoprostatectomy allowed

PATIENT CHARACTERISTICS: Age: Any age Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT no greater than 2 times ULN Renal: Creatinine no greater than 1.7 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: No second degree atrioventricular block or bundle branch block Other: No history of prior malignancy in the past 5 years except basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix No active infection requiring antibiotics No history of allergic reaction to drugs utilizing the vehicle Cremophor Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Recovered from all prior therapies Biologic therapy: No prior biologic response modifier therapy No filgrastim (G-CSF) 24 hours pre- or post-chemotherapy administration Chemotherapy: No prior systemic chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy as a component of bladder sparing therapy No prior adjuvant radiotherapy for locally advanced disease with positive margins Surgery: See Disease Characteristics Other: Prior intravesical therapy for superficial bladder cancer allowed and recovered

Ages: 0 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 490 (Estimated)
Dates: Start 1999-04-02 (Actual); Primary Completion 2001-08 (Actual); Study Completion 2007-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce J. Roth, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (13):
- United States (13):
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Indiana University Hospitals, Indianapolis, Indiana
  - Hunterdon Regional Cancer Center, Flemington, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - South Jersey Hospital - Millville, Millville, New Jersey
  - Fox Chase Cancer Center at Virtua-Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Riverview Medical Center, Red Bank, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Veterans Affairs Medical Center - New York, New York, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Vanderbilt Cancer Center, Nashville, Tennessee